CLINICAL TRIAL: NCT05721651
Title: Efficacy and Safety of Fruquintinib in Combination With PD-1 Inhibitors as First-line Maintenance Therapy for Advanced HER-2 Negative Gastric Cancer: a Single-arm, Prospective, Exploratory Clinical Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wu Jun (Other)
Responsible Party: Sponsor-Investigator, Wu Jun, professor, The First People's Hospital of Changzhou
Organization: The First People's Hospital of Changzhou (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-E2-GC-102
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Fruquintinib+PD-1
  Interventions: Drug: Fruquintinib+PD-1

INTERVENTIONS:
Drug: Fruquintinib+PD-1 — This is a one-arm, prospective, exploratory clinical study, including patients with advanced HER-2-negative gastric cancer (including gastroesophageal junction adenocarcinoma) who received first-line immunization combined with standard chemotherapy (RECIST 1.1 criteria) and were treated with fruquintinib（4mg orally, once daily for 3 wks on/1 wk off ）combined with PD-1 antibody. Until the investigator assesses loss of clinical benefit, unacceptable toxicity, decision by the investigator or subject to withdraw treatment, or death, whichever comes first.
  PD-1: Nivolumab(360mg IV d1, Q3W）；Sintilimab(200mg IV d1, Q3W）；Tislelizumab(200mg IV d1, Q3W） can be selected;

SUMMARY:
Maintenance therapy is very important in advanced HER-2 negative gastric cancer, and immune monotherapy has no obvious benefit in the first-line maintenance treatment of advanced gastric cancer； Fruquintinib is a potent small-molecule VEGFR inhibitor with high kinase selectivity；Studies have shown that immunotherapy combined with antiangiogenic agents is promising for synergistic antitumor effects； The aim of this study was to observe and evaluate the efficacy and safety of Fruquintinib combined with PD-1 inhibitor in the first-line maintenance treatment of advanced HER-2 negative gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, regardless of gender, volunteer to participate in the trial and sign informed consent；
2. Advanced gastric adenocarcinoma confirmed by pathology (including gastroesophageal junction adenocarcinoma) with extragastric measurable lesions (RECIST 1.1 criteria)；
3. Advanced HER-2-negative gastric cancer patients who received first-line PD-1 inhibitors (nivolumab/sindilizumab/tirelizumab) combined with standard chemotherapy and were assessed as non-PD according to RECIST 1.1 criteria；Chemotherapy regimen: SOX/FOLFOX/CAPEOX or fluorouracil combined with purple shirt；Patients receiving single-agent chemotherapy were allowed to enroll；Chemotherapy regimens are used for 4-8 cycles；
4. ECOG score: 0-1；
5. Expect to survive for at least 3 months；
6. Major organ function within 7 days before treatment meets the following criteria: (1) hemoglobin (HB) ≥90 g/L； (2) Absolute neutrophil ANC ≥1.5×109/L； (3) Platelet (PLT) ≥100×109/L；
7. Biochemical tests should meet the following criteria: (1) Total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN), or ≤2.5 times the upper limit of normal value (ULN) in the case of liver metastasis (2) alanine aminotransferase (ALT) and aspartate aminotransferase AST≤2.5 ×ULN, if accompanied by liver metastasis, ALT and AST≤5×ULN(3) Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr)≥60ml/min；
8. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ the lower limit of normal (50%)；
9. Patients of childbearing age (including female and female partners of male patients) must take effective birth control measures
10. he subjects volunteered to participate in this study and signed the ICF；
11. Good compliance is expected, and the efficacy and adverse reactions can be followed up according to the protocol requirements.

Exclusion Criteria:

1. Previous use of antiangiogenic drugs, such as bevacizumab, apatinib, anlotinib, lenvatinib and other antiangiogenic drugs
2. Previous treatment with more than one immune checkpoint inhibitor；
3. Patients who had previously interrupted treatment due to immune-related toxicity during immunotherapy；
4. Patients with severe history of allergy or allergic constitution；
5. Pregnant or lactating women；
6. Patients who have participated in other clinical trials and have not terminated the trial；
7. Patients with a definite propensity for gastrointestinal bleeding. Including the following conditions: ① local active ulcer lesions, and stool occult blood 2+ or abovePatients with fecal occult blood 2+ allowed to retest fecal occult blood and determined by the investigator to have a clear benefit could be enrolled) ② Patients with melena and hematemesis within 3 months； ③ Gastroscopy is required for patients with fecal occult blood 1+ and primary gastric tumor that has not been surgically resected, such as ulcerated gastric cancer, and major gastrointestinal bleeding may occur according to the main investigator of the center；
8. Patients with any severe and/or uncontrolled disease, including: (1) patients with poorly controlled blood pressure (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg)； (2) Patients with grade I or higher myocardial ischemia or infarction, arrhythmias (including QTc ≥ 480ms), or congestive heart failure grade 2 (New York Heart Association (NYHA) classification)； (3) Active or uncontrolled severe infection (≥CTC AE grade 2 infection)； (4) Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis need antiviral therapy； (5) Renal failure requiring hemodialysis or peritoneal dialysis； (6) Have a history of immunodeficiency, including being HIV positive or suffering from other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation； (7) Two consecutive routine urine tests indicated urinary protein ≥++, and confirmed 24-hour urinary protein quantity > 1.0 g； (8) suffer from mental illness, including epilepsy, dementia, severe depression, mania, etc
9. Receiving major surgical treatment, open biopsy or obvious traumatic injury within 28 days before grouping (body-body clinical evaluation)
10. Any history of active autoimmune disease or autoimmune disease, including but not limited to interstitial pneumonia, uveitis, inflammatory bowel disease, hepatitis, pituitary inflammation, vasculitis, systemic lupus erythematosus, etc.
11. Patients whose imaging showed that the tumor had invaded the periphery of important blood vessels or who were judged by the investigator to be highly likely to invade important blood vessels during the subsequent study and cause fatal massive bleeding；
12. Patients with any evidence of bleeding constitution or history, regardless of severity；Patients who had any bleeding or bleeding events ≥CTCAE grade 3 in the 4 weeks before enrollment had unhealed wounds, ulcers, or fractures；
13. 6 months have experienced an arteriovenous thrombotic event, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism；
14. Patients with brain metastases associated with symptoms or symptom control for less than 2 months；
15. Persons with a history of psychotropic drug abuse and inability to abstain or mental disorders；
16. Subjects with dysphagia or known drug absorption disorders；
17. Other conditions deemed inappropriate for inclusion by the investigator。

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 8 weeks, until the occurrence of progressive disease (PD), using RECIST v 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | from randomization until death due to any cause, assessed up to 3 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Objective response rate (ORR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Disease control rate (DCR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Tumor assessment will be performed using radiography method every 8 weeks until the occurrence of progressive disease (PD), using RECIST v 1.1
Safety and tolerance evaluated by incidence, severity and outcomes of AEs | from first dose to 30 days post the last dose
  Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Changzhou, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No